CLINICAL TRIAL: NCT01207947
Title: LEVITRA® Specific Drug Use Investigation. To Investigate the Safety Profile in Combination Use With Alpha-blockers
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13931; LV0702JP (Other: Company internal)
Record Dates: First submitted 2010-09-20; First posted 2010-09-23 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Erectile Dysfunction
Keywords: Vardenafil; Erectile dysfunction; Phosphodiesterase Inhibitors; Combination use with alpha-blockers
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Vardenafil (Levitra, BAY38-9456)

INTERVENTIONS:
Drug: Vardenafil (Levitra, BAY38-9456) — Patients under daily life treatment receiving Levitra according to local drug information.

SUMMARY:
Main object is to investigate the safety profile of Levitra in combination use with alpha-blockers in patients with erectile dysfunction used in clinical practice after launch.

In the initial combination date and the first and second observation after initial combination date, number of tablets prescribed, dose of tablets and number of tablets taken until follow-up visit will be investigated. The efficacy and tolerability will be evaluated at 2 months after initial combination date.

ELIGIBILITY:
Inclusion Criteria:

* Patients >/= 18 years
* Enrollment within 7 days after initiation of combination use of Levitra and alpha-blockers

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Erectile dysfunction patients of 18 years-old or older and also the patients with combination use of alpha-blockers.
Sampling Method: Non-Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of Levitra treatment, namely satisfactory or not is evaluated by inquiring to the enrolled patient according to the following rating scale: 1.very satisfied, 2.satisfied, 3.unsatisfied | 2 months
Safety of Levitra treatment, namely incidence of Adverse Events or Adverse Drug Reactions are evaluated | 2 months

SECONDARY OUTCOMES:
Tolerability of patients with Levitra treatment, namely satisfactory or not is evaluated by inquiring to the enrolled patient according to the following rating scale: 1.very satisfied, 2.satisfied, 3.unsatisfied | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan